CLINICAL TRIAL: NCT02834845
Title: Comparison of Effects of Sevoflurane and Desflurane on Cerebral Oxygenation During Controlled Hypotension
Brief Title: Comparison of Volatile Anesthetics on Cerebral Oxygenation During Controlled Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Perihan Ekmekçi, Associate Professor, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2016Sept
Record Dates: First submitted 2016-06-24; First posted 2016-07-15 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Oxygen Saturation
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental)
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental)
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane %2-3 for general anesthesia maintenance
  Arms: Sevoflurane
Drug: Desflurane — Desflurane %6-8 for general anesthesia maintenance
  Arms: Desflurane

SUMMARY:
Controlled hypotension is a preferred method for reducing surgical bleeding during septoplasty operations however, the level of hypotension and bradycardia should not disrupt cerebral oxygenation. On this account, the investigators aim to investigate the effects of different volatile anesthetics combined with a short-acting opioid on cerebral oxygenation during controlled hypotension using near infrared spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients in American Society of Anesthesiology (ASA) classification I and II
* Patients undergoing elective septoplasty operation

Exclusion Criteria:

* Patients in ASA classification III and higher
* Emergency surgery
* Patients in New York Heart Association classification III-IV
* Patients with known allergy to drugs used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation as measured by Near Infrared Spectroscopy | Duration of surgery
  The effect of sevoflurane and desflurane on NIRS values

SECONDARY OUTCOMES:
Total remifentanil consumption as measured in micrograms | Duration of surgery
The effect of anesthetics on hemodynamic variables | Duration of surgery
  The effects of sevoflurane and desflurane on mean arterial pressure
The effect of anesthetics on hemodynamic variables | Duration of surgery
  The effects of sevoflurane and desflurane on heart rate
The effect of anesthetics on hemodynamic variables | Duration of surgery
  The effects of sevoflurane and desflurane on bispectral index

CONTACTS AND LOCATIONS:
Overall Officials: Ülkü C Köksoy, MD, Principal Investigator — Fellow
Locations (1):
- Ufuk University Hospital, Ankara, Turkey (Türkiye)